CLINICAL TRIAL: NCT00858507
Title: Engaging Homeless Veterans in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 07-184
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Homeless Persons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personal Health Assessment/RN Brief Intervention (Experimental): RN-based medical outreach, administration of a personal health assessment and brief intervention
  Interventions: Behavioral: RN Brief Intervention
- Social Work-Administered Outreach (Placebo Comparator): Social work based outreach (usual care)
  Interventions: Behavioral: Social Worker Outreach

INTERVENTIONS:
Behavioral: RN Brief Intervention — RN administered personal health assessment along with a brief intervention for behavior change administered to homeless veterans in the community
  Arms: Personal Health Assessment/RN Brief Intervention
Behavioral: Social Worker Outreach — Social worker will encounter homeless veteran in the community and encourage to come to the VA for care
  Arms: Social Work-Administered Outreach

SUMMARY:
The objectives of this study are to test an evidence-based model for improving primary and preventive care engagement among homeless Veterans not currently receiving care and to demonstrate the additive benefit of primary care-based treatment engagement by this population.

DETAILED DESCRIPTION:
One out of three homeless men and nearly one quarter of all homeless adults are Veterans. This translates to almost 200,000 Veterans being homeless on any given night. The Department of Veteran Affairs (VA) is a major service provider to homeless persons and has developed several very successful and innovative programs that have been effective in securing housing, economic stability and needed services for these men and women. However, despite these efforts in many communities, Veterans are not accessing these services despite aggressive outreach and state-of-the art programming. The investigators are conducting a prospective randomized controlled trial to test the hypothesis that a personalized health assessment linked to community outreach is more likely to both engage the homeless Veteran in a primary care based chronic disease management model and to sustain that care and associated behavior changes necessary to exit homelessness. The key questions to be addressed in this study are: (1) Will a community-based health-oriented outreach increase health seeking behavior in the intervention group?; (2) can initial engagement be sustained in a continuity care model in this population?; (3) will this intervention facilitate changes/improvements in health seeking behavior that include participation in substance abuse treatment care, compliance with mental health care, and enrollment in VA-based employment/financial support programs?; and (4) can this intervention impact chronic disease management of key cardiovascular risk indicators that disproportionately affect homeless persons?; and (5) do any observed changes correlate with serial behavioral measures and qualitative assessments?

The investigators' working hypothesis is that a targeted outreach to homeless persons that capitalizes on either established or newly realized physical health concerns to affect both health seeking behavior and sustained behavior change. It is grounded in two complementary behavioral models: the Behavioral Model for Vulnerable Populations and the body of research describing intrinsic versus extrinsic motivators for sustained behavior change.

Two hundred and eighty homeless Veterans will be randomized to receive either a personalized health assessment based outreach or usual care (social work/housing focused) outreach. Baseline assessments will include demographics, medical, mental health and substance use co-morbidities, pre-intervention health seeking behavior, readiness for behavior change (URICA), motivation for health care. Serial assessments at months 1, and 6 will assess evolving readiness and motivation as well as changes in their homeless status (sheltering, employment/income, etc.) Actual utilization of services will be assessed using the CPRS electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* VA eligible
* currently homeless

Exclusion Criteria:

* cognitively impaired
* not planning on staying in area for next 6 months
* currently enrolled in VA primary care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P O'Toole, MD, Principal Investigator — VA Medical Center, Providence
Locations (1):
- VA Medical Center, Providence, Providence, Rhode Island, United States

REFERENCES:
- [Result] O'Toole TP, Buckel L, Bourgault C, Blumen J, Redihan SG, Jiang L, Friedmann P. Applying the chronic care model to homeless veterans: effect of a population approach to primary care on utilization and clinical outcomes. Am J Public Health. 2010 Dec;100(12):2493-9. doi: 10.2105/AJPH.2009.179416. Epub 2010 Oct 21. PMID 20966377
- [Result] O'Toole TP, Pirraglia PA, Dosa D, Bourgault C, Redihan S, O'Toole MB, Blumen J; Primary Care-Special Populations Treatment Team. Building care systems to improve access for high-risk and vulnerable veteran populations. J Gen Intern Med. 2011 Nov;26 Suppl 2(Suppl 2):683-8. doi: 10.1007/s11606-011-1818-2. PMID 21989622
- [Result] O'Toole TP, Johnson EE, Borgia ML, Rose J. Tailoring Outreach Efforts to Increase Primary Care Use Among Homeless Veterans: Results of a Randomized Controlled Trial. J Gen Intern Med. 2015 Jul;30(7):886-98. doi: 10.1007/s11606-015-3193-x. Epub 2015 Feb 12. PMID 25673574
- [Result] O'Toole TP, Pape L. Innovative Efforts to Address Homelessness Among Veterans. N C Med J. 2015 Nov-Dec;76(5):311-4. doi: 10.18043/ncm.76.5.311. PMID 26946863

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: RN-based Medical Outreach, Administration of a Personal: RN-based medical outreach, administration of a personal health assessment and brief intervention
  Personal Health Assessment/brief intervention: RN administered personal health assessment along with a brief intervention for behavior change administered to homeless veterans in the community
- Arm 2: Social Work Based Outreach (Usual Care): Social work based outreach (usual care)
  Social work administered outreach: Social worker will encounter homeless veteran in the community and encourage to come to the VA for care
Period: Overall Study
Arm/Group | Arm 1: RN-based Medical Outreach, Administration of a Personal | Arm 2: Social Work Based Outreach (Usual Care)
Started | 105 | 116
Completed | 83 | 101
Not Completed | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: RN-based Medical Outreach, Administration of a Personal | Arm 2: Social Work Based Outreach (Usual Care) | Total
Number analyzed (Participants) | 83 | 101 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 79 | 97 | 176
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.6) | 48.5 (10.2) | 48.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 77 | 97 | 174
Region of Enrollment [Number; unit: participants]
  United States | 83 | 101 | 184

OUTCOME MEASURES:

1. Primary Outcome: Receipt of Primary Care at the VA
Description: The primary aim of this study was to conduct a randomized controlled trial of different interventions aimed at increasing rates of treatment engagement among a community sample of treatment-naive homeless veterans.
Time Frame: within 4 weeks of intervention
Measure: Number; unit: participants
Groups:
- Arm 1: Outreach: RN-based medical outreach, administration of a personal health assessment and brief intervention
  Personal Health Assessment/brief intervention: RN administered personal health assessment along with a brief intervention for behavior change administered to homeless veterans in the community
- Arm 2: Usual Care: Social work based outreach (usual care)
  Social work administered outreach: Social worker will encounter homeless veteran in the community and encourage to come to the VA for care
Arm/Group | Arm 1: Outreach | Arm 2: Usual Care
Number analyzed (Participants) | 83 | 101
participants | 50 | 39

ADVERSE EVENTS:
Description: Per IRB designation as 'minimal risk' and approval of safety monitoring plan, non-serious AEs were not assessed. Serious Adverse Events were not monitored/assessed.
Arm/Group | Arm 1: Outreach | Arm 2: Usual Care
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes